CLINICAL TRIAL: NCT03346928
Title: Free Flaps for Head and Neck Reconstruction : Should we Propose Them to the Elderly
Brief Title: Free Flaps : Should we Propose Them to the Elderly ?
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2017_003
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Head and neck reconstruction — Head and neck free flap reconstruction

SUMMARY:
The objective was to evaluate perioperative morbidity after head and neck microsurgical reconstruction.

DETAILED DESCRIPTION:
The objective was to evaluate perioperative morbidity after head and neck microsurgical reconstruction. A retrospective chart review of all patients undergoing head and neck free flap reconstruction was conducted and the overall hospital length of stay and the incidence of perioperative medical and surgical complications were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer
* Microsurgical free flap reconstruction
* 18 years of age or older

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck cancer undergoing microsurgical free flap reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Medical complications | One month post-surgery
  Occurrence of medical complications within one month post-surgery

SECONDARY OUTCOMES:
Surgical complications | One month post-surgery
  Occurrence of surgical complications within one month post-surgery
Hospital length of stay | Approximately 20 days

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France